CLINICAL TRIAL: NCT02462824
Title: HOme-based moNitORed Exercise for PAD: The HONOR Study
Brief Title: Patient Centered Home Exercise Program for Peripheral Artery Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, Mary McDermott, Jeremiah Stamler Professor in Medicine-General Internal Medicine and Geriatrics and Preventive Medicine, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STU00100697
Record Dates: First submitted 2015-05-04; First posted 2015-06-04 (Estimated); Last update posted 2018-01-08 (Actual); Status verified 2018-01

CONDITIONS: Peripheral Artery Disease
Keywords: Peripheral Artery Disease; Peripheral Arterial Disease; PAD
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Home-based exercise intervention (Experimental): PAD Participants randomized to the home-based exercise intervention will be asked to take part in walking exercise to determine whether a patient-centered home-based exercise program improves walking ability, mobility, pain, and social functioning.
  Interventions: Behavioral: Home-based exercise intervention
- Usual care group (No Intervention): PAD participants randomized to usual care will not receive any study interventions. Rather, they will receive usual care from their own physicians.

INTERVENTIONS:
Behavioral: Home-based exercise intervention — The home-based exercise intervention focuses on walking exercise and consists of two phases. Phase I (weeks 1-4) consists of four on-site visits to an exercise facility, where participants will meet the telephone coach, learn to use the Fitbit activity monitor, become familiar with the study website, learn behavioral skills necessary for long-term adherence to home-based exercise, and get started on their exercise program. Phase II (weeks 5-36) is entirely home-based and includes a) use of the Fitbit for self-monitoring; and b) regularly scheduled telephone calls from the study telephone coach to monitor and support participants' home exercise activity' c) use of the study website; d) optional group telephone calls.
  Arms: Home-based exercise intervention

SUMMARY:
The purpose of this study is to determine the effects of a home-based exercise intervention on walking ability in people with peripheral artery disease. In 200 patients with peripheral artery disease (PAD), the investigators are conducting a randomized controlled trial to determine whether a patient-centered home-based exercise program improves walking ability, physical activity, mobility, pain, and social functioning, compared to a usual care group.

DETAILED DESCRIPTION:
Lower extremity peripheral artery disease (PAD) is a common and chronic condition that affects 8 million people in the United States. PAD patients have difficulty walking because cholesterol blockages in their leg arteries prevent adequate oxygen supply to leg muscles during that activity. PAD patients reduce their physical activity levels and slow their walking speed to avoid leg pain.

Few therapies are available to help PAD patients improve their walking limitations. Treadmill exercise programs that require three or more supervised exercise sessions per week at an exercise facility can help PAD patients walk with less pain. However, most people with PAD do not participate in supervised exercise programs because they are not paid for by medical insurance and the requirements are burdensome for the patients.

The investigators have engaged PAD patients and relevant stakeholders to develop a home-based exercise intervention that is tailored to the needs of the patients. Our home-based exercise intervention includes a Fitbit activity monitor and a coach who will telephone PAD participants at regularly scheduled intervals. PAD patients will use the Fitbit to help them monitor their exercise behavior. The coach will use well-established behavioral methods during the scheduled telephone calls to help PAD patients adhere to regular walking exercise.

The investigators will conduct a randomized controlled trial of 200 patients with PAD to determine whether our home-based walking exercise program significantly improves walking performance and other patient-centered outcomes at the nine-month follow-up, compared to usual care.

PAD patients selected the trial's outcome measures as those that best represent PAD patients' physical limitations. All outcomes are well-validated and accepted outcome measures. The primary outcome measure is the six-minute walk test, an objective measure of walking endurance. Secondary outcomes consist of the Walking Impairment Questionnaire and the PROMIS questionnaires that assess patient-perceived walking ability, mobility, pain, and social functioning.

If our home-based exercise intervention is successful, the intervention will have a substantial impact on the large and growing number of people disabled by PAD.

ELIGIBILITY:
Inclusion Criteria:

1. Participants with an ankle brachial index (ABI) ≤ 0.90 will be eligible for participation.
2. Participants with an ABI > 0.90 but ≤ 1.00 who experience a 20% drop in ankle pressure after the heel-rise exercise will be eligible.
3. Participants with an ABI > 0.90 who have medical record evidence of prior lower extremity revascularization for PAD will be eligible
4. Participants with an ABI > 0.90 who have medical record evidence of PAD based on non-invasive vascular laboratory testing or based on angiographic findings will be eligible. Non-invasive vascular laboratory evidence of PAD must be obtained from a vascular laboratory.

Exclusion Criteria:

1. Above or below knee amputation, critical limb ischemia, wheelchair confinement, foot ulcer, non-English speaking, significant visual impairment that interferes with walking activity, hearing impairment that interferes with full study participation, unable to return to the medical center or fitness center at the expected visit frequency, or unwilling to use technology required for the intervention.
2. Individuals whose walking is limited by a condition other than PAD.
3. Greater than class II NYHA heart failure or angina. Increase in angina, angina at rest, abnormal baseline stress test.
4. Major surgery including lower extremity revascularization or orthopedic surgery during the prior three months or anticipated in the next nine months.
5. Major medical illness including lung disease requiring oxygen, Parkinson's disease that impairs walking ability, or cancer requiring treatment in the prior two years (potential participants may still qualify if they were diagnosed with non-melanoma skin cancer in the past two years or if they have had treatment for an early stage cancer in the past two years and the prognosis is excellent).
6. Heart attack, stroke, or coronary artery bypass surgery in the last 3 months.
7. Mini-mental status examination score < 23, dementia, or psychiatric illness.
8. Currently walking regularly for exercise at a level comparable to the amount of exercise prescribed in the intervention
9. Currently enrolled in another clinical trial, exercise trial, or in cardiac rehabilitation. Currently enrolled in a clinical trial or current participation in cardiac rehabilitation or a trial of a therapeutic intervention within the past three months. For a clinical trial of a stem cell or gene therapy intervention, potential participants will be potentially eligible immediately after the final study visit for the clinical trial, so long as s at least six months has passed since the participant received their final treatment in the stem cell or gene therapy study .
10. Deemed a poor candidate for the study or poorly suited for the intervention (at PI discretion).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2015-04; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Change in Six-Minute Walk Performance at 9-month follow-up | change from baseline to month 9
  In the six-minute walk, participants walk back and forth along a 100-ft hallway for six minutes after standardized instructions to complete as many laps as possible. Distance covered in six minutes is recorded.

SECONDARY OUTCOMES:
Change in Walking Impairment Questionnaire (WIQ) distance and speed and stair-climbing scores between baseline and nine-month follow-up | change from baseline to month 9 follow-up
  The WIQ is a well validated questionnaire that measures patient-reported walking limitations in distance and speed.
Patient-Reported Outcomes Measurement Information System (PROMIS) Questionnaires | change from baseline to month 9 follow-up
  PROMIS Physical Function, PROMIS Pain Interference and PROMIS Ability to Participate in Social Roles and Activities questionnaires will be used to assess patient-reported health status for physical, mental, and social well-being.
Short-Form 36 (SF-36) physical functioning score | change from baseline to month 9 follow-up
  The SF-36 physical functioning score is a well-validated quality of life measure frequently used to assess changes in response to therapeutic interventions in patients with PAD.
Actigraph-measured physical activity. | change in physical activity from baseline to 9 month follow-up
  The Actigraph will be used to measure physical activity.

OTHER OUTCOMES:
Change in Six-Minute Walk Performance at 4.5-month follow-up | change from baseline to month 4.5 follow-up
  In the six-minute walk, participants walk back and forth along a 100-ft hallway for six minutes after standardized instructions to complete as many laps as possible. Distance covered in six minutes is recorded.
Change in Walking Impairment Questionnaire (WIQ) distance and speed and stair-climbing scores between baseline and 4.5 month follow-up | change from baseline to month 4.5 follow-up
  The WIQ is a well validated questionnaire that measures patient-reported walking limitations in distance and speed.
Patient-Reported Outcomes Measurement Information System (PROMIS) Questionnaires | change from baseline to month 4.5 follow-up
  PROMIS Physical Function, PROMIS Pain Interference and PROMIS Ability to Participate in Social Roles and Activities questionnaires will be used to assess patient-reported health status for physical, mental, and social well-being.
Short-Form 36 (SF-36) physical functioning score | change from baseline to month 4.5 follow-up
  The SF-36 physical functioning score is a well-validated quality of life measure frequently used to assess changes in response to therapeutic interventions in patients with PAD.
Actigraph-measured physical activity. | change in physical activity from baseline to 4.5 month follow-up
  The Actigraph will be used to measure physical activity.

CONTACTS AND LOCATIONS:
Overall Officials: Mary McDermott, MD, Principal Investigator — Northwestern University
Locations (4):
- United States (4):
  - Northwestern University Feinberg School of Medicine, Chicago, Illinois
  - Northwestern University feinberg School of Medicine, Chicago, Illinois
  - University of Minnesota, Minneapolis, Minnesota
  - New York University School of Medicine, New York, New York

REFERENCES:
- [Derived] McDermott MM, Spring B, Berger JS, Treat-Jacobson D, Conte MS, Creager MA, Criqui MH, Ferrucci L, Gornik HL, Guralnik JM, Hahn EA, Henke P, Kibbe MR, Kohlman-Trighoff D, Li L, Lloyd-Jones D, McCarthy W, Polonsky TS, Skelly C, Tian L, Zhao L, Zhang D, Rejeski WJ. Effect of a Home-Based Exercise Intervention of Wearable Technology and Telephone Coaching on Walking Performance in Peripheral Artery Disease: The HONOR Randomized Clinical Trial. JAMA. 2018 Apr 24;319(16):1665-1676. doi: 10.1001/jama.2018.3275. PMID 29710165